CLINICAL TRIAL: NCT04417283
Title: Project HOPE 1000: A Longitudinal Study of Mothers and Infants to Understand Health Outcomes Related to Pregnancy and Early-Life Exposures
Brief Title: Project HOPE 1000: Health Outcomes Pregnancy Exposures
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00100000
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Pregnant
Keywords: Pregnancy; Gestation; Placenta; Exposure; Environment; Social Drivers of Health; Infancy; Biological specimens; Electronic health records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mother-infant dyads: Mother and/or infant participants will provide a series of biological specimens, including blood, urine, and microbiome samples. Additionally, each participant will wear a silicone wrist band each trimester to capture environmental exposures and will fill out study surveys related to diet, environmental exposures, and social factors.

SUMMARY:
The purpose of this study is to collect biological samples from pregnant women and their babies and to collect data on long-term health, school outcomes, and the use of state and county services. The information learned from this study may help identify important factors that may influence the health of mothers and babies, both short-and long-term.

DETAILED DESCRIPTION:
Humans pass through more biological milestones during gestation and the first two years of life (known as the "first 1000 days") than during any other period of development. Consequently, both intrinsic biology/physiology and extrinsic factors such as environmental exposures can have profound impacts on long-term health and disease outcomes. The purpose of this project is to develop a cohort of mother-infant dyads that can provide a collection of birth samples and be studied long-term - from pregnancy through early childhood - to help identify early life factors that influence lifelong health and disease. The study will include collection of specimens from pregnant women during each trimester of pregnancy, at delivery, and within the first few months after giving birth, as well as collection of specimens from the infants at birth and during their first two years of life. In addition to specimens, health information will be collected from the participants' electronic health records, and via questionnaires to assess health behaviors, social determinants, and environmental exposures. Participants may also consent for yearly review of state administrative data, including educational data, social services, and vital records. The specimens and data collected in this study will allow for assessment of the impact of different factors during pregnancy and early childhood on long-term health and well-being.

ELIGIBILITY:
Inclusion criteria:

* The subject has provided a signed Informed consent prior to any study procedures.
* Maternal age at consent of ≥ 18 years old
* Ability to understand English or Spanish
* Willingness to comply with and be available for all protocol procedures
* Singleton gestation < 24 weeks 0 days
* Receiving prenatal care at a Duke-affiliated Obstetrics clinic with the intent of delivering at Duke University Health System-affiliated hospital (including Duke University Hospital and Duke Regional Hospital)
* Plans to have their infant seen at a Duke-affiliated Pediatrics practice after birth
* Plans to remain in the area for two years after delivery

Exclusion criteria:

* Non-viable pregnancy
* Having any condition that, in the opinion of the site investigators, would place the subject at unacceptable risk of injury or confound data interpretation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant participants can enroll in the first or second trimester of pregnancy
Study Population: Mother and/or infant participants will provide a series of biological specimens, including blood, urine, and microbiome samples. Additionally, each participant will wear a silicone wrist band each trimester to capture environmental exposures and will fill out study surveys related to diet, environmental exposures, and social factors.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Development of a data repository to provide a secure, centralized storage location for samples from pregnant women. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gilner, MD, Principal Investigator — Duke University
Locations (1):
- Duke affiliated ObGyn clinics within Duke Health, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No